CLINICAL TRIAL: NCT05495698
Title: Triple Therapy Convenience by the Use of One or Multiple Inhalers and Digital Support in Chronic Obstructive Pulmonary Disease
Acronym: TRICOLON
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Franciscus Gasthuis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: FranciscusGasthuis
Record Dates: First submitted 2022-08-05; First posted 2022-08-10 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Copd; Adherence, Medication
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Medication Adherence | interventions — Beclomethasone

STUDY DESIGN:
Intervention Model Description: The first group will receive multi-inhaler triple therapy (control group), the second group single inhaler triple therapy (intervention group 1) and the third group single inhaler triple therapy with extra digital support to increase therapy adherence (intervention group 2).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control group (Other): multi-inhaler triple therapy (Qvar and Bevespi)
  Interventions: Drug: multi-inhaler triple therapy (Qvar + Bevespi)
- Intervention group 1 (Other): single-inhaler triple therapy (Trimbow)
  Interventions: Drug: single-inhaler triple therapy (Trimbow)
- Intervention group 2 (Other): single-inhaler triple therapy (Trimbow) + e-health applications
  Interventions: Drug: single-inhaler triple therapy (Trimbow); Device: E-health application: Curavista app & FindAir e-device

INTERVENTIONS:
Drug: single-inhaler triple therapy (Trimbow) — Patients in the intervention group will receive the triple therapy in one inhaler in stead of multiple inhalers. The actual medication is the same.
  Arms: Intervention group 1; Intervention group 2
Device: E-health application: Curavista app & FindAir e-device — Patients in intervention group 2 will receive Trimbow and will use the health app of Curavista and the smart-inhaler of FindAir
  Arms: Intervention group 2
Drug: multi-inhaler triple therapy (Qvar + Bevespi) — Patients in the intervention group will receive the triple therapy in multiple inhalers. The actual medication is the same.
  Arms: Control group

SUMMARY:
TRICOLON is an investigator initiated, prospective, interventional, open-label, randomized, real-world, multi-centre, 3-arms study in the Netherlands. The primary objective is to investigate in COPD patients if single-inhaler triple therapy (SITT) is superior to multi-inhaler triple therapy (MITT) in terms of adherence to inhaled corticosteroids (ICS) therapy and to investigate if SITT with e-health support is superior to MITT and SITT without e-health support.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of COPD for at least 1 year before the screening visit
* Aged 40 years and older
* An indication for triple therapy according to the treating physician (following the GOLD guideline 2021(2)). Could be step-up from dual therapy or currently receiving triple therapy (both MITT and SITT).
* Owner of mobile device compatible with e-device app with access to internet (Android or iOS)
* Willing to provide written informed consent
* Current or ex-smoker

Exclusion Criteria:

* Inability to comply with study procedures or with study treatment
* Insufficiently skilled in the Dutch language to be able to read and understand the app. Help by third party (family members) is allowed
* Asthma as the predominant disease according to the investigator's opinion, a past history of asthma is allowed
* Use of e-health application for COPD in the past six months
* Patients with any other therapy that could interfere with the study drugs (according to the investigator's opinion)
* Use of nebulized bronchodilators, for example via pari boy
* Pregnant or lactating women and all women physiologically capable of becoming pregnant unless they have highly effective contraceptive
* Patients mentally or legally incapacitated, or patients accommodated in an establishment as a result of an official or judicial order
* Patients without the capability to complete the questionnaires

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2022-12-13 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Adherence to ICS therapy | 12 months
  average adherence to ICS therapy (expressed as a percentage, measured as the number of actuations registered by the e-device divided by the total number of prescribed doses) over 12 months of treatment

SECONDARY OUTCOMES:
TAI questionnaire score | 12 months
  questionnaire that identifies non-adherence and gives insight in the barriers related to the use of inhalers in asthma and COPD
CCQ questionnaire | 12 months
  measures health status and can be used to assess health-related quality of life
VAS score | 12 months
  a non-specific scale to score an outcome from 0 (not satisfied at all) to 10 (extremely satisfied)
PIH-NL | 12 months
  12-item scale to measure self-management behaviour and knowledge of patients with chronic diseases as COPD
WPAI | 12 months
  questionnaire to measure impairments in work and activities
EQ-5D-5L | 12 months
  questionnaire to assess the health-status
HLS-EU-Q16 | 12 months
  assessment of patients' health literacy
Number exacerbations | 12 months
  A moderate exacerbation is defined as sustained worsening of the patient's condition, from a stable state and beyond day-to-day variation, that is acute in onset and warrants additional treatment (systemic corticosteroids and/or antibiotics). An exacerbation is defined as severe if hospitalization or emergency department visit is necessary
SABA use | 12 months
  Use of espace medication

OTHER OUTCOMES:
Concentration of beclomethasone and formoterol in hair | 2-3 months
  In a subgroup of patients, beclomethasone and formoterol concentration in their hair will be measured

CONTACTS AND LOCATIONS:
Locations (1):
- Franciscus Gasthuis & Vlietland, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Cuperus LJA, van der Palen J, Aldenkamp A, van Huisstede A, Bischoff EWMA, van Boven JFM, Brijker F, Dik S, van Excel JAJM, Goosens M, van Hal PTW, Kuijvenhoven JC, Kunz LIZ, Vasbinder EC, Kerstjens HAM, In 't Veen JCCM; TRICOLON study group. Adherence to single inhaler triple therapy and digital inhalers in Chronic Obstructive Pulmonary Disease: a literature review and protocol for a randomized controlled trial (TRICOLON study). BMC Pulm Med. 2024 Jul 4;24(1):317. doi: 10.1186/s12890-024-03044-3. PMID 38965541